CLINICAL TRIAL: NCT02921113
Title: Soluble Urokinase Plasminogen Activator Receptor (suPAR) in the Early Diagnosis of Acute Kidney Injury After On-Pump Cardiac Surgery
Brief Title: suPAR in the Early Diagnosis of Acute Kidney Injury(AKI) After On-Pump Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2016.236
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Acute Kidney Injury
Keywords: suPAR; Acute Kidney Injury; On-Pump Cardiac Surgery; Biomarker
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma(suPAR) plasma(NGAL) urine NGAL serum creatinine plasma Cystatine C
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute Kidney Injury(AKI) is of the serious complications in patients with undergoing on-pump cardiac surgery. End stage kidney failure requiring dialysis therapy after cardiac surgery is associated with more than 60% mortality rate. Involvement of AKI after on-pump cardiac surgery increases the mortality rate 19 times. suPAR is one of the novel biomarker which has potential prognostic value for renal dysfunction in patients with undergoing on-pump cardiac surgery. Early diagnosis and prompt intervention to prevent AKI has great importance for management of postoperative cardiac patients.

ELIGIBILITY:
Inclusion Criteria:

* Approved informed concent Age higher than 18 years old

Exclusion Criteria:

* Chronic kidney disease Renal transplantation Cancer history Previous cardiac surgery Sepsis Liver failure Thyroid dysfunction Having long term steroid therapy Having renal replacement therapy Exposure to nephrotoxic drug and radiocontrast substance before 5 days of surgery Diagnosis of Acute Kidney Injury Intraaortic balloon or Extracorporeal Membrane Oxygenation insertion after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective on-pump cardiac surgery with no known kidney disease
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | 2 days
  Patients will be classified as AKI patients and non-AKI patients according to KDIGO classification. AKI patients will be subdivided into 3 subgroup according to KDIGO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bünyamin KIR, M.D, Principal Investigator — Marmara University School of Medicine Dept of Anesthesiology and Reanimation; İsmail Cinel, Prof. M.D, Study Director — Marmara University School of Medicine Dept of Anesthesiology and Reanimation; Beliz Bilgili, Asst. Prof., Principal Investigator — Marmara University School of Medicine Dept. of Anesthesiology and Reanimation; Sinan Arsan, Prof. M.D, Principal Investigator — Marmara University School of Medicine Dept. of Cardiovascular Surgery
Locations (1):
- Department of Anesthesiology, Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Khan E, Batuman V, Lertora JJ. Emergence of biomarkers in nephropharmacology. Biomark Med. 2010 Dec;4(6):805-14. doi: 10.2217/bmm.10.115. PMID 21133700
- [Result] Chertow GM, Lazarus JM, Christiansen CL, Cook EF, Hammermeister KE, Grover F, Daley J. Preoperative renal risk stratification. Circulation. 1997 Feb 18;95(4):878-84. doi: 10.1161/01.cir.95.4.878. PMID 9054745
- [Result] Wei C, El Hindi S, Li J, Fornoni A, Goes N, Sageshima J, Maiguel D, Karumanchi SA, Yap HK, Saleem M, Zhang Q, Nikolic B, Chaudhuri A, Daftarian P, Salido E, Torres A, Salifu M, Sarwal MM, Schaefer F, Morath C, Schwenger V, Zeier M, Gupta V, Roth D, Rastaldi MP, Burke G, Ruiz P, Reiser J. Circulating urokinase receptor as a cause of focal segmental glomerulosclerosis. Nat Med. 2011 Jul 31;17(8):952-60. doi: 10.1038/nm.2411. PMID 21804539
- [Result] Jalkanen V, Yang R, Linko R, Huhtala H, Okkonen M, Varpula T, Pettila V, Tenhunen J; FINNALI Study Group. SuPAR and PAI-1 in critically ill, mechanically ventilated patients. Intensive Care Med. 2013 Mar;39(3):489-96. doi: 10.1007/s00134-012-2730-x. Epub 2012 Oct 26. PMID 23100007
- [Result] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219